CLINICAL TRIAL: NCT01923831
Title: Comparison of the Effect of Magnesium Sulfate and Dexamethasone on Postoperative Sore Throat After Spinal Surgery in Prone Position With Tracheal Intubation: a Double-blind, Randomized, Noninferiority Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2013-0385
Record Dates: First submitted 2013-08-05; First posted 2013-08-16 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Post Operative Sore Throat
Keywords: Magnesium, Post operative sore throat, Prone position, Tracheal intubation
MeSH Terms: interventions — Magnesium Sulfate; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium group (Experimental)
  Interventions: Drug: Magnesium Sulfate
- Dexamethasone group (Active Comparator)
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium sulfate 30 mg kg-1 was infused in 100mL normal saline for 10 minutes immediately before anesthesia induction. After tracheal intubation, normal saline 1.6mL ( equivalent volume as Dexamethasone 8mg) was injected, and magnesium sulfate was continuously infused at the rate of 10 mg Kg-1 h-1 until the end of surgery. (at the time of skin closure)
  Arms: Magnesium group
Drug: dexamethasone — Normal saline 100mL was infused for 10 minutes immediately before anesthesia induction. After tracheal intubation, dexamethasone 8mg was injected, and normal saline was continuously infused at the rate of 10 mg Kg-1 h-1 until the end of surgery. (at the time of skin closure)
  Arms: Dexamethasone group

SUMMARY:
The purpose of this study is to compare the effect of magnesium sulfate and dexamethasone on postoperative sore throat after spinal surgery in prone position with tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients aged between 20 and 65 year undergoing 1 or 2 level posterior spinal fusion in prone position with tracheal intubation

Exclusion Criteria:

* preexisting hoarseness or sore throat, upper respiratory tract infection
* steroid therapy or immunocompromised patients
* chronic treatment with calcium channel blocker or magnesium
* allergy to magnesium sulphate
* Cormack-Lehane grade 3,4 or patients who are expected to difficult intubation
* fail to tracheal intubation at first trial
* reduced kidney function
* Diabetes mellitus

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The effect of magnesium sulfate on postoperative sore throat after spinal surgery in prone position with tracheal intubation | Change of post operative sore throat level from 1 to 48 hours after surgery
  Incidence of post operative sore throat Severity of post operative sore throat (10 cm-visual analogue scale ) Incidence of post operative hoarseness Severity of post operative hoarseness ( four-graded scale, 0= no hoarseness, 1= mild hoarseness, 2= severe hoarseness, 3= aphonia)

SECONDARY OUTCOMES:
The effect of dexamethasone on postoperative sore throat after spinal surgery in prone position with tracheal intubation | Change of post operative sore throat level from 1 to 48 hours after surgery
  Incidence of post operative sore throat Severity of post operative sore throat (10 cm-visual analogue scale ) Incidence of post operative hoarseness Severity of post operative hoarseness ( four-graded scale, 0= no hoarseness, 1= mild hoarseness, 2= severe hoarseness, 3= aphonia)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea